CLINICAL TRIAL: NCT00346177
Title: Injection of Autologous CD34+ Cells for Neovascularization and Symptom Relief in Patients With Myocardial Ischemia and LVEF < 40%
Brief Title: Stem Cell Study for Patients With Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding not obtained. No subjects enrolled.
Sponsor: Losordo, Douglas, M.D. (Individual)
Responsible Party: Director, Feinberg Cardiovascular Research Institute, Program in Cardiovascular Regenerative Medicine, Northwestern University/Northwestern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB-IND-11196-02
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Myocardial Ischemia; Congestive Heart Failure; Cardiovascular Disease
Keywords: heart; stem Cells; low EF; heart attack; cardiomyopathy; congestive heart failure; cardiovascular disease; Heart Failure; Low Ejection Fraction
MeSH Terms: conditions — Myocardial Ischemia; Heart Failure; Cardiovascular Diseases; Myocardial Infarction; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Stem Cells
  Interventions: Biological: Autologous Stem Cells
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Autologous Stem Cells

INTERVENTIONS:
Biological: Autologous Stem Cells — Intramyocardial injections

SUMMARY:
The purpose of this study is to determine if cell therapy with your own cells (autologous cells) delivered with a catheter to regions of the heart with poor blood flow will be safe and if it will improve your ejection fraction and heart failure symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than 21 years old.
* Subjects with functional class (NYHA) III ischemic heart failure.
* Subjects who have attempted "best" cardiac medical therapy including long-acting nitrates, maximal use of beta-adrenergic blocking agents, and angiotensin-converting enzyme inhibitors without control of symptoms.
* Subjects must be identified as non-candidates for conventional revascularization by their referring cardiologist. The patient's angiogram will then be reviewed by an independent interventional cardiologist and independent cardiac surgeon to determine if the patient is eligible for revascularization.
* Subjects must have left ventricular ejection fraction <40% by echocardiography.
* All subjects must have a recent coronary angiogram (within the last 1 year) to document the coronary anatomy and insure the presence of coronary disease that is not amenable to standard revascularization procedures.
* Have serum B-type Natriuretic Peptide (BNP) level >100 pg/ml.

Exclusion Criteria:

* Myocardial infarction (Q wave or non-Q wave defined as CKMB >3 times normal) within 30 days of treatment.
* Successful coronary revascularization procedures within 3 months of study enrollment.
* Documented stroke or transient ischemic attack (TIA) within 60 days of study enrollment.
* NYHA Class I, II or IV heart failure and patients with idiopathic or non-ischemic heart failure.
* History of severe aortic stenosis (aortic valve area < 1.0 cm2) or insufficiency (>2+); severe mitral stenosis (mitral valve area <1.5 cm2); or severe mitral insufficiency(>2+).
* Implantation of biventricular pacemaker within 90 days of study treatment.
* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year, such as chronic medical illness (i.e. severe chronic obstructive pulmonary disease, renal failure or cancer).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
The purpose of this study is to determine if cell therapy with your own cells (autologous cells) delivered with a catheter to regions of the heart with poor blood flow will be safe and if it will improve your ejection fraction and heart failure symptoms. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Losordo, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States